CLINICAL TRIAL: NCT03454152
Title: Electrocardiogram and Echocardiography Changes in Children With Diabetic Ketoacidosis
Brief Title: Ecg & Echo Changes in Children With DKA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatima Younis, Principal investigator, Assiut University
Other Study IDs: DKA2018
Record Dates: First submitted 2018-02-18; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Pediatric Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: pediatric patients with diabetic ketoacidosis come to Assuit University Children Hospital within one year. Electrocardiogram and echocardiography will be done to all patient with diabetic ketoacidosis

SUMMARY:
Diabetic ketoacidosis (DKA) is an important complication of childhood diabetes mellitus and the most frequent diabetes-related cause of death in children.

Diabetic ketoacidosis (DKA) is caused by a decrease in effective circulating insulin associated with increases in counter regulatory hormones including glucagon, catecholamines, cortisol, and growth hormone. This leads to increased glucose production by the liver and kidney and impaired peripheral glucose utilisation with resultant hyperglycaemia, and hyperosmolality. Increased lipolysis, with ketone body (beta-hydroxybutyrate, acetoacetate) production causes ketonaemia and metabolic acidosis. Hyperglycaemia and acidosis result in osmotic diuresis, dehydration, and obligate loss of electrolytes.

DETAILED DESCRIPTION:
DKA can affect cardiovascular function through several mechanisms. The effect of acidosis on the heart depends upon the pH level. In mild acidosis, there is increased catecholamine release which is compensated by increased inotropy, chronotropy, cardiac output and peripheral vascular resistance. When acidosis is severe, i.e. pH is less than 7.2, the H+ ions have a direct cardiac depressant action.

Fluid and electrolyte imbalance is very common in DKA, Potassium deficit is one of the most important of electrolyte imbalances seen in DKA as it can lead to fatal arrhythmias. The most common and perhaps the earliest ECG finding in hypokalemia is a prominent U wave, usually evident in leads II and III. The most common cardiac arrhythmias are atrial premature contractions, atrial tachycardia with or without atrioventricular block, supraventricular and ventricular premature contractions.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged : 1 month -18years with diabetic ketoacidosis

Exclusion Criteria:

* Pediatric Patients who have associated cardiovascular disease. ( congenital or rheumatic).
* Pediatric patients with hyperglycemic hyperosmolar state.
* Pediatric patients with other causes of metabolic acidosis.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients with diabetic ketoacidosis come to Assuit University Children Hospital within one year.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Echocardiography parameters | baseline
  Right and left ventricular dimension during diabetic ketoacidosis and after correction.
Electrocardiogram parameters | baseline
  QT interval and PR interval.

SECONDARY OUTCOMES:
Electrocardiogram changes | baseline
  ST segment elevation or depression
Echocardiography findings | baseline
  Systolic and diastolic left ventricular function

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edge JA, Ford-Adams ME, Dunger DB. Causes of death in children with insulin dependent diabetes 1990-96. Arch Dis Child. 1999 Oct;81(4):318-23. doi: 10.1136/adc.81.4.318. PMID 10490436
- [Background] Dunger DB, Sperling MA, Acerini CL, Bohn DJ, Daneman D, Danne TP, Glaser NS, Hanas R, Hintz RL, Levitsky LL, Savage MO, Tasker RC, Wolfsdorf JI; ESPE; LWPES. ESPE/LWPES consensus statement on diabetic ketoacidosis in children and adolescents. Arch Dis Child. 2004 Feb;89(2):188-94. doi: 10.1136/adc.2003.044875. PMID 14736641
- [Background] Gandhi MJ, Suvarna TT. Cardiovascular complications in diabetic ketoacidosis. Int J Diab Dev Countries. 1995;15:132-133.
- [Background] Chung EK. Electrolyte imbalance and cardiac arrhythmias. In : Principles of Cardiac Arrhythmias. Edward Chung (ed.) Williams and Wilkins, 1989.